CLINICAL TRIAL: NCT06042062
Title: Clinical Evaluation of Infection Control to Knee Periprosthetic Joint Infection (PJI) -United Cellbrick Knee Spacer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: United Orthopedic Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202300966A3
Record Dates: First submitted 2023-08-14; First posted 2023-09-18 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2023-08

CONDITIONS: Knee; Infection, Joint
Keywords: Infection Control; Two-Stage Exchange Arthroplasty; Knee Spacer
MeSH Terms: conditions — Infections | interventions — Metered Dose Inhalers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "Spacer" group (Experimental): The subjects who are assigned to Articulating Spacers in two-stage exchange arthroplasty.
  Interventions: Device: Spacer
- "Novel spacer" group (Experimental): The subjects who are assigned to United Cellbrick Knee Spacer in two-stage exchange arthroplasty.
  Interventions: Device: Novel spacer

INTERVENTIONS:
Device: Novel spacer — After diagnosis of infection and informed consent, patients will be taken to the operating room. After anesthetization, patients will be randomized to either a United Cellbrick spacer (United Orthopedic Corporation, Taiwan) or an articulating full-cement spacer. Randomization will be performed by prepared opaque envelopes administered by a nonparticipant in the study. After a complete debridement of devitalized tissue, explantation of the infected components and any associated cement, either a Cellbrick spacer or an articulating spacer will be placed. As for the United Cellbrick spacer, antibiotic loaded bone cement (ALBC) will be molded into the designed holes (fenestrations). The ALBC will be formed from an antibiotic mixture of Vancomycin and Gentamicin with bone cement (Stryker, Simplex P).
  Arms: "Novel spacer" group
Device: Spacer — After diagnosis of infection and informed consent, patients will be taken to the operating room. After anesthetization, patients will be randomized to either a Cellbrick spacer (United Orthopedic Corporation, Taiwan) or an articulating full-cement spacer. Randomization will be performed by prepared opaque envelopes administered by a nonparticipant in the study. After a complete debridement of devitalized tissue, explantation of the infected components and any associated cement, either an United Cellbrick spacer or an Articulating Spacer will be placed. The Articulating Spacer will be hand-made to fit the femoral and tibial exposed metaphyses as a solid block with associated antibiotic loaded bone cement (ALBC). The ALBC will be formed from an antibiotic mixture of Vancomycin and Gentamicin with bone cement (Stryker, Simplex P).
  Arms: "Spacer" group

SUMMARY:
A novel polyethylene-based knee spacer (United Cellbrick Knee Spacer), for the purpose of infection control, was developed to enhance biomechanical safety and surgical convenience of articulating knee spacers. In the present study, Articulating Spacers were compared to the United Cellbrick Knee Spacers in a practical setting to enhance our understanding of the safety and performance of United Cellbrick Knee Spacer.

DETAILED DESCRIPTION:
Two-stage exchange arthroplasty, which involves the removal of infected prostheses and introduction of a temporary antibiotic-loaded cement spacers at the infection site, has been widely accepted among treatment options. Antibiotic-loaded cement spacers facilitate in maintaining joint space, limb length, soft tissue tension, and lengthening the period of effective antibiotic release until infection control has been accomplished.

Although articulating knee spacers have demonstrated advantages in joint mobility and clinically successful rates in infection control, issues relating to biomechanical safety contributed by cement material characteristics have been noted. Surgeons had to implement alternative methods for the construction of an intramedullary spacer to provide sufficient infection control for deeper infection sites which could cause surgical inconveniences. A novel polyethylene-based knee spacer, for the purpose of infection control, was developed to enhance biomechanical safety and surgical convenience of articulating knee spacers.

The investigators aim to conduct a clinical study comparing the use of Articulating Spacers to United Cellbrick Knee Spacers in a practical setting to better understand the safety and performance of United Cellbrick Knee Spacers and to enhance the clinical confidence of investigators. A total of 10 participants who are undergoing two-stage exchange arthroplasty at Linkou Changgung Memorial Hospital will be recruited, including 5 participants in the "Spacer" group and 5 participants in the "Novel Spacer" group.

Participants in the "Spacer" group will receive a full-cement spacer (Stryker, Simplex P) made of broad-acting antibiotics (Vancomycin and Gentamicin) produced in the hospital.

Participants in the "Novel Spacer" group will receive a United Cellbrick Knee Spacer, where the femoral and tibial spacers will be filled with bone cement (Stryker Simplex P) with antibiotics (Vancomycin and Gentamicin).

Spacer survivorship defined as no removal or revision of any components as a result of mechanical failure or complications will be analyzed. Blood tests, joint effusions, and x-ray inspections will also be collected for analysis.

ELIGIBILITY:
Inclusion Criteria

Patients who are 18 years of age or older, suitable for temporary knee joint implants, and will be undergoing treatment in Linkou Chang Gung Memorial Hospital who meet the following criteria and have skeletally mature bones:

1. Patients who are diagnosed with infection before surgery and are expected to undergo two-stage procedure for total knee replacement (TKR);
2. Patients who are willing to use traditional mobility aids (such as crutches, walkers) during implantation;
3. The implantation time of the temporary knee implant shall not exceed 180 days.

Exclusion Criteria

1. Patients who are allergic to or have suffered from allergies to any component of the implant, the bone cement used together or antibiotics.
2. Patients who cannot perform two-stage knee replacement surgery due to decreased immune response or other relevant clinical conditions.
3. Patients who have not previously received total knee replacement surgery, and the secondary infection is caused by trauma, septic arthritis or other surgery.
4. Sufficient support and / or fixation for implants due to disease, soft tissue defects, bone defects or other relevant clinical conditions.
5. Inability or unwillingness to return to hospital for evaluation.
6. Cognitive function impairment makes the subject unable to answer questions or cooperate with instructions.
7. Other systemic comorbidities lead to severe impairment of the subject's mobility and function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Success Rate | up to 6 months following surgery
  Failure is defined as removal or revision of any components as a result of mechanical failure or complications.
  Success is defined as implants that are successfully implanted without any failure for the duration of up to 180 days.
  *Note: Spacers are temporarily implanted into patients for any two-stage arthroplasty. Hence, upon assessment by the surgeon, when the condition of the patients are ideal for the second-stage arthroplasty procedure, the surgeon will remove the spacer accordingly. Therefore, the timeframe for the spacer removal may happen anywhere before the duration of 180 days.
  The success rate will be represented as a percentage (%).

SECONDARY OUTCOMES:
Vancomycin Concentration | Day 1, 3, 7, up to 6 months following surgery
  Vancomycin Concentration will be quantified utilizing Particle Enhanced Turbidimetric Inhibition Immunoassay. Blood samples (3mL) and joint effusion samples (5-10cc) will both be used to analyze the efficacy of vancomycin concentration (5-15ug/mL).
Gentamycin Concentration | Day 1, 3, 7, up to 6 months following surgery
  Gentamycin Concentration will be quantified utilizing Particle Enhanced Turbidimetric Inhibition Immunoassay. Blood samples (3mL) and joint effusion samples (5-10cc) will both be used to analyze the efficacy of gentamycin concentration (5-15ug/mL).
C-reactive protein assessment | Baseline, 7, up to 6 months following surgery
  C-reactive protein assessment will be quantified utilizing turbidimetric-immunoassay. Blood samples (3mL) will be used to determine the level of inflammation.
Bioassay of Antibiotic Activity of in Vitro Samples | Day 1, 2, 3, 7
  Bioassay of Antibiotic Activity of in Vitro Samples will be quantified utilizing aliquots of the samples and a modified microtube dilution bioassay. The following strains were selected as test organisms: Methicillin-susceptible Staphylococcus aureus (MSSA, ATCC 25923), Methicillin-resistant Staphylococcus aureus (MRSA, ATCC 43300), Staphylococcus epidermidis (ATCC 14990), Pseudomonas aeruginosa (P. aeruginosa, ATCC 27853) or Escherichia coli (E. coli, ATCC 25922). The in vitro samples were were inoculated with 105 colony forming units (CFUs) of bacteria per milliliter in 96-well culture dishes and incubated at 37 degree Celsius for 24 hours according to Hsu et al. The growth of bacteria associated with the different concentrations of antibiotics was compared visibly with each other and against the positive control (without antibiotic). The minimum inhibitory concentration of each antibiotic against each bacterium was determined by microtube dilution bioassay.
Spacer Complications | Baseline, Day 0, up to 6 months following surgery
  Any issues with spacer complications including allergic reactions, bone loss, joint stiffness, wound complications, recurrence or persistence of the infection, spacer fracture or dislocation, and side effects of local or systemic antibiotics will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Han Chang, MD, PhD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Department of Orthopedic Surgery at Linkou Changgung Memorial Hospital, Taoyuan District, Taiwan